CLINICAL TRIAL: NCT05142423
Title: An Open Label, Multi-center, Phase Ib/II Clinical Study of AK109 Combined With AK104 to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity in Advanced Solid Tumors
Brief Title: A Study of AK109 Combined With AK104 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK109-102
Record Dates: First submitted 2021-10-29; First posted 2021-12-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK109+AK104 (Experimental): AK104: 10mg/kg (d1, q3w); AK109: 10mg/kg or 15mg/kg(d1, q3w)
  Interventions: Drug: AK109+AK104

INTERVENTIONS:
Drug: AK109+AK104 — It includes dose escalation and dose expansion stage. 6-12 patients will be enrolled in dose escalation stage for safety and efficacy. Then select specific dose of AK104 and AK109. Expand for the further safety and efficacy study.

SUMMARY:
This is a multi-center, open label, phase Ib/II clinical study of AK109 and AK104 to evaluate the safety, tolerability, effectiveness, pharmacokinetic characteristics in advanced solid tumors .

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Age ≥ 18 years and ≤ 75 years.
3. ECOG Performance Status of 0 or 1.
4. Estimated life expectancy of ≥3 months.
5. Histologically or cytologically documented, locally advanced or metastatic solid tumours (NSCLC, mCRC, HCC, GEJ, etc. ), for which standard therapy does not exist or has proven ineffective or intolerable.
6. At least one radiographically measurable lesion per RECIST 1.1.
7. Tumor biopsy (during advanced stage) available.
8. Adequate organ function.
9. Female participants of childbearing potential and male partners with female partners of childbearing potential must agree to use effective barrier methods of contraception during the study and for 120 days after last dose of study drug.

Exclusion Criteria:

1. Other documented active malignancies other than for this trial within 3 years.
2. Participation in other clincial trials simultaneously.
3. Use of systemic anti-tumor treatments with 4 weeks, non-specific immunomodulating agents within 2 weeks.
4. Prior exposure to other T cell coregulatory proteins except for PD-1/PD-L1 inhibitors (apart from cohort B, i.e. treatment naive HCC patients).
5. Current use corticosteroids/immunosuppressive agents, permanently discontinuation of study drug, or having any unresolved irAEs (≥grade 2) from prior PD-1/PD-L1 inhibitors treatment.
6. Central nervous system (CNS) metastasis, meningeal metastasis, spinal cord compression, or leptomeningeal disease.
7. Uncontrolled pleural/pericardial or peritoneal effusion.
8. History of hemorrhagic event need blood transfusion, invasive approaches to intervene, or hospitalization within 3 months, or having high risks of bleeding.
9. Any thromboembolic event, non-gastrointestinal fistula or female genital tract fistula within 6 months.
10. Uncontrolled gastrointestinal diseases.
11. Use of NSAIDs and anticoagulant agents within 7 days.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks.
13. Severe or uncontrolled hypertension and cardiovascular/cerebrovascular diseases.
14. Uncontrolled comorbidities need corticosteroids using.
15. Active or prior autoimmune disease or history of immunodeficiency.
16. History of interstitial lung disease.
17. Known history of active tuberculosis (TB).
18. Evidence of active infections including hepatitis B and C.
19. Use of anti-infectious agents within 2 weeks.
20. History of human immunodeficiency virus (HIV) infections.
21. Active syphilis infections.
22. Any unresolved toxicities (≥grade 2) from previous anti-cancer therapies.
23. Mental illness, drug abuse, or alcohol dependence that may affect compliance with the test requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing dose-limiting toxicities(DLTs) | Up to 21 days
  DLTs will be assessed during the first 21 days of treatment and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications.
Incidences and severity of AE | Up to 2 years
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with CR or PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1) or death from any cause (whichever occurs first)
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to 2 years
  Time to response (TTR) is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR, as determined by the investigator according to RECIST v1.1.
Overall survival (OS) | Up to 2 years
  OS defined as the time from the first dose to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Correlation analysis of PD-L1 expression with efficacy | Up to 2 years
  Characteristics of tumor tissue PD-L1 expression and exploratory analysis of correlation between PD-L1 expression status and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Nong Xu, MD, Principal Investigator — The First Affiliated Hospital of Medicine College, Zhejiang University; Jianming Xu, MD, Principal Investigator — The Chinese PLA General Hospital
Locations (1):
- First affliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No